CLINICAL TRIAL: NCT01648023
Title: Comparative, Prospective, Open-labeled, Randomized Phase II Study of Cisplatin or Carboplatin With Gemcitabine in Combination With Irinotecan-loaded Beads (LC or ONCOZENE) Versus Cisplatin or Carboplatin With Gemcitabine Alone in the Treatment of Patients With Unresectable Intrahepatic Cholangiocarcinoma
Brief Title: Drug-Eluting Bead, Irinotecan Therapy for Unresectable Intrahepatic Cholangiocarcinoma w/Concomitant Gemcitabine and Cisplatin or Carboplatin
Acronym: DELTIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robert C. Martin (Other)
Responsible Party: Sponsor-Investigator, Robert C. Martin, Professor, University of Louisville
Organization: University of Louisville (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-0181
Record Dates: First submitted 2012-07-17; First posted 2012-07-24 (Estimated); Results first posted 2022-01-13 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2021-12

CONDITIONS: Unresectable Intrahepatic Cholangiocarcinoma
Keywords: LC Bead; Irinotecan; ONCOZENE BEAD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Randomization to LC OR ONCOZENE Bead with Gem-Cis or Gem-Carbo (Experimental): Transarterial Chemoembolization (LC or ONCOZENE Bead) with Gem-Cis or Gem-Carbo
  Interventions: Device: LC or ONCOZENE Bead with Gem-Cis or Gem-Carbo
- Randomization to Gem-Cis or Gem-Carbo (Active Comparator): Gem-Cis or Gem-Carbo alone
  Interventions: Drug: Gem-Cis or Gem-Carbo

INTERVENTIONS:
Device: LC or ONCOZENE Bead with Gem-Cis or Gem-Carbo
  Arms: Randomization to LC OR ONCOZENE Bead with Gem-Cis or Gem-Carbo
Drug: Gem-Cis or Gem-Carbo
  Arms: Randomization to Gem-Cis or Gem-Carbo

SUMMARY:
The purpose of this study is to find out if the combination of trans-arterial chemoembolization (LC or ONCOZENE BEAD) plus infusional chemotherapy is safe and more effective than just receiving the infusional chemotherapy alone.

ELIGIBILITY:
Inclusion:

* Patients over 18 years of age, of any race or sex, who have histologic and radiologic evidence of intrahepatic cholangiocarcinoma, who have been deemed unresectable by an experienced hepatic surgeon, and who are able to give informed consent, will be eligible
* Patients with at least one measurable liver tumor, with size > 1cm (modified RECIST criteria)
* Patients with liver-dominant disease defined as ≥80% tumor burden confined to the liver
* Non-pregnant with an acceptable contraception in premenopausal women.
* Hematologic function: ANC ≥ 1.5 x 109/L, platelets ≥ 75 x109/L, INR ≤1.3 (patients on therapeutic anticoagulants are not eligible if they can not stop there anti-coagulation prior to DEBIRI and meet INR criteria)
* Adequate liver function as measured by: Total bilirubin ≤ 2.0 mg/dl,
* Adequate renal function (creatinine ≤ 2.3 mg/dl)
* Women of child bearing potential and fertile men are required to use effective contraception (negative serum βHCG for women of child-bearing age)
* Signed, written informed consent
* Less than 70% of liver parenchymal tumor replacement

Exclusion:

* Patient eligible for curative treatment (i.e. resection or tumor ablation).
* Active bacterial, viral or fungal infection within 72 hours of study entry
* Women who are pregnant or breast feeding
* ECOG Performance Status score of >3
* Life expectancy of < 3 months
* Allergy to contrast media that cannot be managed with standard care (e.g. steroids), making magnetic resonance imaging (MRI) or computed tomography (CT) contraindicated
* Presence of another malignancy with the exception of cervical carcinoma in situ and stage I basal or squamous cell carcinoma of the skin.
* Any contraindication for hepatic embolization procedures:
* Large shunt as determined by the investigator (pretesting with TcMMA not required)
* Severe atheromatosis vascular disease that precludes arterial cannulization
* Hepatofugal blood flow
* Main portal vein occlusion (e.g. thrombus or tumor)
* Other significant medical or surgical condition, or any medication or treatment, that would place the patient at undue risk and that would preclude the safe use of chemoembolization or would interfere with study participation
* Patients with prior contraindications for the use of irinotecan, gemcitabine, or cisplatin
* Patients who have received prior systemic therapy with either irinotecan, gemcitabine, or cisplatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-07; Primary Completion 2019-01 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Martin, MD, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Randomization to LC OR ONCOZENE Bead With Gem-Cis or Gem-Carbo: Transarterial Chemoembolization (LC or ONCOZENE Bead) with Gem-Cis or Gem-Carbo
  LC or ONCOZENE Bead with Gem-Cis or Gem-Carbo
- Randomization to Gem-Cis or Gem-Carbo: Gem-Cis or Gem-Carbo alone
  Gem-Cis or Gem-Carbo
Period: Overall Study
Arm/Group | Randomization to LC OR ONCOZENE Bead With Gem-Cis or Gem-Carbo | Randomization to Gem-Cis or Gem-Carbo
Started | 25 | 24
Completed | 24 | 22
Not Completed | 1 | 2
Not completed — Screen Fail Post Randomization | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomization to LC OR ONCOZENE Bead With Gem-Cis or Gem-Carbo | Randomization to Gem-Cis or Gem-Carbo | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 13 | 28
  >=65 years | 9 | 9 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 11 | 9 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 21 | 19 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response (Overall Response = Complete Response + Partial Response + Progressive Disease + Stable Disease)
Description: Tumor response will be determined using Modified Response Evaluation Criteria in Solid Tumors (mRECIST). Response will be classified as: Complete Response - disappearance of all lesions; Partial Response - at least 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of the longest diameter or 30% reduction in arterial enhancement; Progressive Disease - at least 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest longest diameter recorded since start of treatment or appearance of one or more new lesions greater than 1cm in size; Stable Disease - neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum longest diameter since start of treatment.
Time Frame: Assessed at 2, 4 and 6 months. 6 months reported.
Measure: Number; unit: participants
Arm/Group | Randomization to LC OR ONCOZENE Bead With Gem-Cis or Gem-Carbo | Randomization to Gem-Cis or Gem-Carbo
Number analyzed (Participants) | 24 | 22
participants | 24 | 22

2. Secondary Outcome: Overall Survival
Description: Long-term follow-up will occur every 3-4 months for up to one year after discontinuation of active study treatment. Subjects who have completed the long-term follow-up period will be monitored every 3 - 6 months until evidence of progression of disease. Once there is progression of disease subjects will be followed for overall survival by telephone or standard physician follow-ups as per standard of care until death.
Time Frame: 4.5 Years
Population: All randomized subjects who receive at least one cycle of intravenous chemotherapy or LC or ONCOZENE beads loaded with irinotecan. Subjects will be grouped according to their randomization.
Measure: Median (Full Range); unit: Months
Arm/Group | Randomization to LC OR ONCOZENE Bead With Gem-Cis or Gem-Carbo | Randomization to Gem-Cis or Gem-Carbo
Number analyzed (Participants) | 24 | 22
Months | 33.7 [13.5 to 54.5] | 12.6 [8.7 to 33.4]

ADVERSE EVENTS:
Time Frame: Adverse and Serious Adverse Events were assessed for 15 months. All-Cause Morality was assessed from randomization to Date of Death from Any Cause (up to 55 months)
Arm/Group | Randomization to LC OR ONCOZENE Bead With Gem-Cis or Gem-Carbo | Randomization to Gem-Cis or Gem-Carbo
All-Cause Mortality (participants affected / at risk) | 17/24 | 16/22
Serious Adverse Events (participants affected / at risk) | 21/24 | 19/22
Other Adverse Events (participants affected / at risk) | 24/24 | 19/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomization to LC OR ONCOZENE Bead With Gem-Cis or Gem-Carbo (N=24) | Randomization to Gem-Cis or Gem-Carbo (N=22)
Abdominal Pain (Gastrointestinal disorders) | 1 | 2
Acute Cardiac Injury (Cardiac disorders) | 0 | 1
Acute Cardiorespiratory Distress (Cardiac disorders) | 0 | 1
Acute Cholycystitis (Gastrointestinal disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Acute Renal Failure (Renal and urinary disorders) | 1 | 1
Acute Renal Insufficiency (Renal and urinary disorders) | 1 | 0
Acute Small Bowel Obstruction (Gastrointestinal disorders) | 1 | 1
Altered Mental Status (Psychiatric disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0
Biliary Obstruction (Hepatobiliary disorders) | 1 | 0
Biliary Strictures (Hepatobiliary disorders) | 1 | 0
Biliary Tract Infection (Hepatobiliary disorders) | 1 | 0
Congestive Heart Failure (Cardiac disorders) | 1 | 0
Dehydration (General disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Enterocutaneous Fistula (Gastrointestinal disorders) | 0 | 1
ESBL E Coli Bacteremia (Infections and infestations) | 1 | 0
ESBL E Coli Urinary Tract Infection (Infections and infestations) | 1 | 0
Fatigue (General disorders) | 0 | 1
Fever (General disorders) | 2 | 0
Hypercalcemia (Investigations) | 0 | 1
Hypertension (Cardiac disorders) | 2 | 1
Hypoglycemia (Investigations) | 1 | 0
Ischemic Colitis (Gastrointestinal disorders) | 0 | 1
Lethargy (General disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Liver Abscess (Hepatobiliary disorders) | 1 | 1
Liver Failure (Hepatobiliary disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 1
Nausea (General disorders) | 4 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenic Fever (Blood and lymphatic system disorders) | 2 | 0
Neutropenic Sepsis (Infections and infestations) | 2 | 0
Oversedation (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pelvic Fracture (Musculoskeletal and connective tissue disorders) | 0 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 2 | 2
Stroke (Vascular disorders) | 1 | 1
Subarachnoid Hemorrhage (General disorders) | 1 | 0
Subcapsular Liver Abscess (Hepatobiliary disorders) | 1 | 0
Systemic Inflammatory Response Syndrome (General disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
TIA (Vascular disorders) | 1 | 0
Upper GI Hemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Wound Infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomization to LC OR ONCOZENE Bead With Gem-Cis or Gem-Carbo (N=24) | Randomization to Gem-Cis or Gem-Carbo (N=22)
Abdominal Distension (Gastrointestinal disorders) | 3 | 2
Abdominal Pain (Gastrointestinal disorders) | 21 | 5
Gout (Immune system disorders) | 0 | 1
Agitation (General disorders) | 1 | 1
Aguesia (General disorders) | 3 | 0
Alopecia (Immune system disorders) | 3 | 2
Anemia (Blood and lymphatic system disorders) | 12 | 9
Anorexia (General disorders) | 3 | 1
Anxiety (Psychiatric disorders) | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Ascites (Hepatobiliary disorders) | 2 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Balance Problems (General disorders) | 2 | 0
Edema (General disorders) | 7 | 6
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Body Aches (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone Pain (General disorders) | 2 | 1
Bruising (Blood and lymphatic system disorders) | 2 | 2
C Difficile (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Cachexia (General disorders) | 0 | 1
Chills (General disorders) | 3 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cold Sensitivity (General disorders) | 1 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 17 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Decreased Appetite (General disorders) | 5 | 3
Dysgeusia (General disorders) | 2 | 7
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Thrombosis (Blood and lymphatic system disorders) | 3 | 2
Dehydration (General disorders) | 4 | 4
Delirium (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Diaphoresis (General disorders) | 5 | 0
Diarrhea (Gastrointestinal disorders) | 10 | 7
Dizziness (General disorders) | 5 | 3
Dyspenea (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Dyspepsia (Gastrointestinal disorders) | 3 | 2
Dysuria (Renal and urinary disorders) | 1 | 2
Otitis Media (Ear and labyrinth disorders) | 0 | 2
Early Satiety (General disorders) | 2 | 0
Elevated Liver Enzymes (Investigations) | 9 | 3
Encephalopathy (General disorders) | 0 | 1
Epistaxis (Blood and lymphatic system disorders) | 2 | 2
Esophageal Varices (Gastrointestinal disorders) | 0 | 1
Failure to Thrive (General disorders) | 1 | 0
Fall (General disorders) | 2 | 0
Fatigue (General disorders) | 22 | 6
Fecal Incontinence (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 11 | 3
Gait Disturbance (General disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 2 | 1
GERD (Gastrointestinal disorders) | 0 | 1
Headache (General disorders) | 4 | 5
Heartburn (Gastrointestinal disorders) | 2 | 1
Hematemesis (General disorders) | 0 | 1
Hemopthysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperbilirubinemia (Investigations) | 1 | 0
Hypercalcemia (Investigations) | 1 | 1
Hyperglycemia (Investigations) | 4 | 2
Hyperkalemia (Investigations) | 2 | 0
Hypernatremia (Investigations) | 1 | 0
Hypertension (Vascular disorders) | 12 | 1
Hypocalcemia (Investigations) | 1 | 1
Hypokalemia (Investigations) | 4 | 3
Hypomagnesemia (Investigations) | 10 | 6
Hyponatremia (Investigations) | 3 | 0
Hypotension (Vascular disorders) | 2 | 2
Influenza (Infections and infestations) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0
Insomnia (General disorders) | 6 | 1
Ischemic Cardiomyopathy (Cardiac disorders) | 1 | 0
Jaundice (General disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Leukopenia (Investigations) | 6 | 3
Malabsorption (Gastrointestinal disorders) | 0 | 1
Malaise (General disorders) | 1 | 2
Malnutrition (General disorders) | 2 | 2
Pericardial Effusion (Cardiac disorders) | 1 | 0
Mucositis (General disorders) | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 20 | 12
Neutropenia (Investigations) | 8 | 8
Pancytopenia (Blood and lymphatic system disorders) | 2 | 1
Parasthesia (General disorders) | 1 | 1
Peripheral Neuropathy (Nervous system disorders) | 7 | 2
Rash (General disorders) | 3 | 1
Syncope (General disorders) | 3 | 0
Tachycardia (Cardiac disorders) | 4 | 1
Thrombocytopenia (Investigations) | 10 | 7
Upper Respiratory Infection (Infections and infestations) | 4 | 0
Vomiting (Gastrointestinal disorders) | 15 | 6
Urinary Tract Infection (Renal and urinary disorders) | 4 | 4
Weakness (General disorders) | 3 | 3
weight Loss (Gastrointestinal disorders) | 6 | 1
Tremors (General disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT01648023/Prot_SAP_000.pdf